CLINICAL TRIAL: NCT03577444
Title: Role of Genetic Polymorphism in Neuroplasticity Involved in Dysphagia Recovery
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Associate Professor, The Catholic University of Korea
Other Study IDs: NTRH-18001
Record Dates: First submitted 2018-06-08; First posted 2018-07-05 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Stroke; Dysphagia
Keywords: gene polymorphism; stroke; dysphagia; poststroke recovery
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dysphagia patients: Patients who had been diagnosed with neurogenic dysphagia related to either stroke or traumatic brain injury at two university affiliated hospitals

SUMMARY:
The purpose of this study is to assess the association of genetic polymorphism such as the Brain-derived Neurotrophic factor (BDNF), in neurogenic dysphagia in those with brain lesion.

DETAILED DESCRIPTION:
Neurogenic dysphagia attributable to acquired brain lesions, such as after stroke and after traumatic brain injury, are one of leading causes of chronic disability world widely and it is expected to substantially increase over the next two decades. Among various sequalae, dysphagia can be observed in about 40% -60% of post-stroke patients and 20% -30% of them might suffer from recurrent aspiration pneumonia and may inhibit recovery and can even lead to death. Recovery after brain lesions can be explained by specific molecular events. It is proven that Genetic polymorphisms associated with impaired neural repair or plasticity might reduce recovery from stroke. Not only for the motor recovery, but genetic polymorphism is also crucial for the recovery of swallowing after stroke, however, only limited amount of studies are available. Therefore, it is urgent to determine whether the recovery of swallowing disorders after stroke is affected by the inherent polymorphism of the patient, whether the degree of recovery and brain plasticity associated with swallowing depend on the gene characteristics and polymorphism of the patient and whether recovery in swallowing parallel to the recovery observed in other functional areas (ie. hand recovery, truncal control recovery, ADL recovery).

Based on the results of this study, results will be expected to help provide genetically tailored diagnosis and prognostication according to the gene polymorphism of the patient. Optimized treatment of the patient is expected to contribute to prevention of respiratory complications and improve functional outcome related to swallowing after stroke.

ELIGIBILITY:
Inclusion Criteria

1. Patients who had been diagnosed with first ever brain lesions ( stroke and traumatic brain lessons) and referred to Department of Rehabilitation( in Bucheon St. Mary's Hospital and National Traffic Injury Rehabilitation Hospital)
2. Patients who were hospitalized for 30 days and were followed up at 3 months after the onset of brain lesions
3. Patients who agree to participate in the study or if the guardian or legal representative agrees only if the patient has difficulties in consenting or consenting to participate directly in the language disability.
4. In the case of a suspected feeding swallowing disorder in the patient, the patient should be confirmed by VFSS(Videofluoroscopic Swallwing Study) or FEES(Fiberoptic Endoscopic Evaluation of Swallowing)

Exclusion Criteria

1. Patients who do not meet the above criteria
2. Patients with difficulty in collecting blood for genetic testing
3. Patients who were not able to followed-up for 6 months(follow up loss patients)
4. Patients with long-term Parkinson's disease, Alzheimer's disease, Guillain-Barre syndrome, myasthenia gravis syndrome, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had were diagnosed with first dysphagia and referred to Department of Rehabilitation( in Bucheon St. Mary's Hospital and National Traffic Injury Rehabilitation Hospital) with medical records up to 6 months after onset of brain lesion
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2018-08-04 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Change in Functional Oral Intake Scale(FOIS) | initial 4 weeks,3months after onset
  Functional oral intake scale(FOIS) is categorical scale range from 1 indicating severe dysphagia and 7 indicating safe oral feeding. Higher change in FOIS indicates improvement of patient's swallowing function.

SECONDARY OUTCOMES:
Change in Berg Balance Scale(BBS) | initial 4 weeks, 3 months after onset
  BBS is a scale that measure person's static and dynamic balance abilities, ranging from 0 to 56 where 56 indicated independence in gait and 0 means unable to gait. Higher change in Berg Balance Scale means improved patient's mobility.
Change in Medical Research Council(MRC) grade Disability level | initial 4 weeks, 3 months after onset
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  It is categorical value with the the scale running from 0-6, running from perfect health without symptoms to death.
Change in K-MBI(Korean Modified Barthel Index) | initial 4 weeks, 3 months after onset
  The Barthel scale or Barthel ADL index is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. Higher scores indicates indolence in ADL activities.
Change in FAC(Functional Ambulatory Category) | initial 4 weeks, 3 months after onset
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device . Higher scores indicate better performance.
Change in Fugyl Meyer score from baseline | initial 4 weeks, 3 months after onset
  The Fugl-Meyer Assessment for upper extremity (FMA-UE)is considered to assess the body function according to the International Classification of Functioning, Disability and Health (ICF) with a maximum score of 66 points)
Change in MMSE-K(Korean Minimental Status Examination) | initial 4 weeks,3months after onset
  3. The Mini-Mental State Examination (MMSE) is a 30-point questionnaire that is used extensively to measure cognitive impairment.[1] Higher score indicates better cognitive function.
Change in scores of Quality of Life Survey score (EQ5D(EuroQol-5 dimension) | initial 4 weeks, 3months after onset
  The QOLS is a reliable and valid instrument for measuring quality of life from the perspective of the patient The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change in Penetration-Aspiration Scale(PAS) | 4 weeks, 3 months after onset
  initial PAS is a categorical scale that measures level of penetration of bolus(food) into airway at pharynx. It ranges from Score 1 to 8, where 1 indicated no airway entrance of bolus and 8 indicated glottic passage of food. Higher change in PAS indicates improvement in patient's swallowing function.
Change in dysphagia outcome rating scale | 4 weeks, 3 months after onset
  initial The Dysphagia Outcome and Severity Scale (DOSS) is a simple, easy-to-use, 7-point scale developed to systematically rate the functional severity of dysphagia based on objective assessment and make recommendations for diet level, independence level, and type of nutrition with level 1 indicating severe dysphagia and level 7 indicating normal swallowing function.
Change in SWAL-QOL(swallowing quality of life)) survey score | 4 weeks, 3 months after onset
  initial SWAL-QOL is a survey that evaluation patient's subjective quality of life within their swallowing function. Scored will be sumed up where higher score indicates better quality of life.
Number of events associated with aspiration pneumonia | 4 weeks, 3 months after onset
  initial Diagnosis of aspiration pneumonia will be based on ≥3 of the following features: fever (>38°C), productive cough, abnormal respiratory examination, abnormal chest radiograph; specifically involving the dependent portions of the lung; white blood cell count >12,000/mL, or isolation of a relevant pathogen and use of antibiotics)

CONTACTS AND LOCATIONS:
Overall Officials: TaeWoo Kim, Study Director — National Traffic Rehabilitation Hospital Korea
Locations (2):
- South Korea (2):
  - Department of Rehabilitation Medicine, Bucheon-si, Gyonggido
  - Department of Rehabilitation Medicine Bucheon St Mary's Hospital, Catholic University of Korea, College of Medicine, Bucheon-si, Kyounggido

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park HY, Kim Y, Oh HM, Kim TW, Park GY, Im S. Potential Prognostic Impact of Dopamine Receptor D1 (rs4532) Polymorphism in Post-stroke Outcome in the Elderly. Front Neurol. 2021 Jun 30;12:675060. doi: 10.3389/fneur.2021.675060. eCollection 2021. PMID 34276537
- [Derived] Oh HM, Kim TW, Park HY, Kim Y, Park GY, Im S. Role of rs6265 BDNF polymorphisms and post-stroke dysphagia recovery-A prospective cohort study. Neurogastroenterol Motil. 2021 Jan;33(1):e13953. doi: 10.1111/nmo.13953. Epub 2020 Aug 9. PMID 32776402